CLINICAL TRIAL: NCT06791785
Title: The Effect Of Aromatherapy Applied To Children Aged 9-12 On Exam Anxiety, Attention Deficit and Academic Success
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ferhat Gunerigok, LECTURER, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-59090411-44-98875002
Record Dates: First submitted 2024-12-31; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Aromatherapy; Test Anxiety; Attention Deficits; Academic Achievement; Child
Keywords: Child; Test Anxiety; Attention Deficit; Academic Achievement; Aromatherapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lemon (Experimental): For the lemon group, 550 ml of pure water will be poured into the diffusers to be placed in the classroom, and 3 drops of lemon aroma oil will be dropped into the pure water from the aromatherapy oil bottle.
  Interventions: Other: Before Application; Other: Before the 1st Written Exam; Other: End of Term
- Lavender (Experimental): For the lavender group, 550 ml of pure water will be poured into the diffusers to be placed in the classroom, and 3 drops of lavender aroma oil will be dropped into the pure water from the aromatherapy oil bottle.
  Interventions: Other: Before Application; Other: Before the 1st Written Exam; Other: End of Term
- Placebo (Placebo Comparator): For the placebo group, the impression of oil will be given by dropping 3 drops of pure water from an oil bottle with a similar structure but containing pure water.
  Interventions: Other: Before Application; Other: Before the 1st Written Exam; Other: End of Term

INTERVENTIONS:
Other: Before Application — All groups will be asked to fill out forms before the application (Westside test anxiety scale, burdon attention test, descriptive information form)
Other: Before the 1st Written Exam — Fill out forms before the 1st written exam (Westside test anxiety scale, burdon attention test, descriptive information form)
Other: End of Term — Fill out forms at the end of the term (Westside test anxiety scale, burdon attention test, descriptive information form)

SUMMARY:
This study was planned to examine the effects of aromatherapy applied to children aged 9-12 on exam anxiety, attention deficit and academic success. The study was conducted as single blind.

Hypotheses of the Study H1: Children given lemon aroma with an aromatherapy diffuser have higher Burdon Attention Test mean scores than children in the placebo group; H1.1. Burdon Attention Test mean scores are higher. H1.2. Westside Exam Anxiety mean scores are lower. H2: Children given lavender aroma with an aromatherapy diffuser have higher Burdon Attention Test mean scores than children in the placebo group; H2.1. Burdon Attention Test mean scores are higher. H2.2. Westside Exam Anxiety mean scores are lower. H3: Children given lavender aroma with an aromatherapy diffuser have lower Westside Exam Anxiety mean scores than children given lemon aroma; H3.1. Westside Exam Anxiety mean scores are lower. H3.2. Burdon Attention Test mean scores are higher.

DETAILED DESCRIPTION:
Aromatherapy is stated to be based on the therapeutic use of volatile oils obtained from plants and aromatic liquids obtained from the bark and flowers of plants. The liquids used in aromatherapy applications are generally in the form of oil and are very diverse; mint, lemon (citrus limon), laurel, lavender (lavandula angustifolia), eucalyptus, Rumi chamomile, rosemary, tea tree, frankincense, immortelle, fennel, camphor, cypress, pine, tangerine, ginger, grapefruit, etc.

When the application methods are examined, it is stated that they are in the form of gel, body bath, hot towel, facial steam, inhalation (sniffing, dropping on a handkerchief, directly smelling the bottle), steam inhalation.

When the effects of aromatherapy oils are examined in the literature; It is stated that it has many effects such as anxiety and stress reliever, antioxidant, beneficial for menstrual pain, sedative, immune supporter, anti-inflammatory, antimicrobial, antispasmodic, antitussive (cough suppressant), decongestant, febrifuge (fever reducer), mucolytic (expectorant), mourning and sadness reliever, detoxifier, vasoconstrictor, analgesic, antiemetic, carminative (inhibitor and elimination of intestinal gases, facilitating digestion). When the effects of lemon oil (citrus limon oil) and lavender (lavandula angustifolia) oil to be used in this research are examined; lavender (lavandula angustifolia): calming, anxiety reliever, wound repairer, healing properties in burns, cell regenerator, itching reducer and ideal effects for children; lemon oil has stress-relieving properties, increases energy, supports immunity and has antimicrobial effects. When looking at the mechanism of action of aromatherapy on humans, it is stated that it triggers the release of substances such as dopamine, serotonin, endorphin and noradrenaline in the cerebellum and causes changes in the person's mental and physical state. When the use of aromatherapy oils throughout history is examined, it is seen that it was first used in the ancient Egyptian civilization in the making of mummies and in the ancient Chinese civilization as an expression of gratitude to God. It is stated that the use of aromatherapy for therapeutic and beauty purposes first emerged in ancient Greek civilizations. It is stated that during the Roman Empire, aromatherapy was used with massage techniques after baths. When looking at its first use in nursing, it is stated that it started with Florence Nightingale and that she tried to relax patients who were suffering during the war by applying lavender oil to their foreheads. Aromatherapy, which also has a long history in nursing care, is stated to be one of the methods that nurses can use to improve patient care and strengthen nursing. It is stated that nursing is a dynamic profession and that when the information in the literature changes, this change is quickly adapted to and that it is important for them to use this change and improve themselves in the areas they work in (school health, community health, child health, etc.). Aromatherapy applications are one of these variables used in different ages and different educational areas in the literature.

This study is planned to be conducted due to the limited number of studies on inhalation aromatherapy as an intervention in the context of neurocognitive anxiety, stress, memory and attention, intelligence, academic performance, etc. in the context of school health within the scope of a holistic approach in the child population and the need for nursing studies in this area. The preadolescent period selected in this study is stated to be the period between the ages of 9-12, known as the period when many physical and psychological changes occur. Therefore, this study aims to evaluate the effects of aromatherapy on exam anxiety, attention deficit and academic success of 9-12 year old children in the school age group. It is thought that the results will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 9-12
* Must have family permission to participate in the study
* Must have children who can give consent to participate in the study

Exclusion Criteria:

* Having a chronic disease related to the respiratory system
* Being allergic to lemon or lavender aroma
* Being a child with special needs
* Being included in an Individualized Education Program (IEP)
* Developing any problems during the application

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Power Analysis and Time | It will take approximately 4-4.5 months until the spring semester education is completed.
  Input Parameters:
  * Effect size (f): 0.5 (A medium-high effect size)
  * α error prob: 0.05 (Type I error rate, 5%)
  * Power (1-β err prob): 0.95 (Power, 95%)
  * Number of groups: 3 (Number of groups)
  Output Parameters:
  * Noncentrality parameter λ: 16.5
  * Critical F: 3.14281 (Critical F value for ANOVA)
  * Numerator df (degrees of freedom): 2 (Groups - 1)
  * Denominator df: 63 (Sample size - number of groups)
  * Total sample size: 66 (Calculated total sample size)
  * Actual power: 0.95347 (Quite close to the expected power)
  Accuracy of Calculations:
  * It is seen that an analysis suitable for the input values was performed.
  * The total sample size (66) is reasonable given the given α, power, and effect size.
  If you plan to run an ANOVA test with these parameters, the results will be valid. A total sample size of 66 is sufficient for 3 groups.
  TİME: It will take approximately 4-4.5 months until the spring semester education is completed.
Data Analysis and G*Power Analysis | It will take approximately 4-4.5 months until the spring semester education is completed.
  The survey and scale data to be obtained will be analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Mean, standard deviation, median, minimum and maximum values will be used in the descriptive statistics of the data. Kurtosis and skewness values of the distributions will be examined in order to determine whether the distributions show a normal distribution in determining the statistical techniques to be used in the analysis of the data. The relationship between the three variables will be examined with the One Way Anova Test. Chi-Square analysis will be applied while examining the relationships between the groups of nominal variables. In order to determine whether the difference between the test score averages before the application, after the 1st written exam and at the end of the term is significant between the groups, variance analysis will be applied in repeated measurements (one-way for group and time, two-way for group*time).

CONTACTS AND LOCATIONS:
Locations (1):
- Güzeltepe Ortaokulu, Istanbul, Eyüpsultan, Turkey (Türkiye)